CLINICAL TRIAL: NCT05445752
Title: Conservative Nodal Surgery (Node-picking) of Patients With Stage III Melanoma With Low-burden of Nodal Disease (MELCONSURG MULTICENTRE COHORT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Other Study IDs: MELCONSURG
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Melanoma Stage III
Keywords: Surgery; Lymph node dissection; Conservative nodal surgery; Lymph node metastasis; Melanoma; Stage III melanoma
MeSH Terms: conditions — Melanoma; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Standard treatment for stage III melanoma with lymph node metastases involves complete lymph node dissection, which is a radical surgical procedure aimed at the removal of the entire regional lymph node basin. Conservative surgery for low-burden nodal metastasis involves removal of the metastatic lymph node or nodes ("node-picking"), leaving uninvolved nodes within the regional basin. This is expected to provide adequate regional control of the disease with no negative impact on patient survival and a lower rate of surgical complications.

Aims: The MelConSurg Cohort will provide the first data on conservative surgery for patients with stage III melanoma with nodal metastases detected clinically or by imaging.

Methods: A multicentre, single-arm prospective cohort study. Inclusion criteria: Patients with melanoma aged between 18 and 90 years, Eastern Cooperative Oncology Group performance status 0-1, non-matted regional lymph node metastasis (N1b or N2b) in a single regional basin detected clinically or by imaging (ultrasound, CT scan, PET scan). Study period: A 3-year recruitment period and a 3-year follow-up phase.

Intervention: Patients will undergo conservative nodal surgery using conventional surgery, radio-guided surgery, or imaging guided surgery.

Outcome measures: 3-year nodal relapse-free survival, 3-year disease-free survival, 3-year melanoma-specific survival, rate of surgical complications, and quality of life (SF-36 questionnaire).

Sample size & Statistics: the estimated sample size to be recruited is 68 patients. Survival outcomes will be analysed through the Kaplan-Meier method, with the log-rank test. Conclusions: This Project is expected to provide unique evidence regarding a less radical nodal surgery for patients with melanoma. If favourable results are obtained, controlled studies could be conducted and changes in current clinical practice could be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with melanoma aged between 18 and 90 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Nodal stage N1b or N2b (American Joint Committee on Cancer 8th edition) in a single regional basin detected clinically or by imaging (ultrasound, CT scan, PET scan).

Exclusion Criteria:

* Single lymph node metastasis in more than one regional basin.
* Multiple primary melanoma (except for limb melanoma).
* Primary occult melanoma.
* Previous nodal, locoregional, or distant metastasis.
* Previous lymph node surgery, except for SLNB.
* Distant metastases detected at the screening evaluations or first postoperative PET-CT scan.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Melanoma patients (stage III N1b or N2b) fulfilling inclusion criteria and with no exclusion criteria managed at any of the participant centers.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Nodal relapse-free survival | 3-year
  The primary outcome measure is the frequency and time to develop recurrence in the same nodal basin.

SECONDARY OUTCOMES:
Disease-free survival | 3-year
  Frequency and time to develop recurrence at any site, both regional or at distance.
Melanoma-specific survival | 3-year
  Frequency and time to death directly related to melanoma progression.
Surgical complication rate | 3-year
  Frequency of long-term complications (seroma, lymphedema, nerve injury, others). health-related quality of life questionnaire.
Quality of life | 3-year
  Quality of life as tested by the SF-36 health-related quality of life questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Department. University Hospital Virgen Macarena, Seville, Spain